CLINICAL TRIAL: NCT04918420
Title: Efficacy and Safety of the Flow Diverter (Tonbridge) for Endovascular Treatment of Intracranial Aneurysms: A Prospective, Multi-center, Single-arm Trial
Brief Title: A Single-arm Trial of the Flow Diverter (Tonbridge) For Endovascular Treatment of Intracranial Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ton-Bridge Medical Tech. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZHTQ2021002
Record Dates: First submitted 2021-05-31; First posted 2021-06-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flow Diverter (Tonbridge) (Experimental): Treatment with Flow Diverter (Tonbridge)
  Interventions: Device: Flow Diverter (Tonbridge)

INTERVENTIONS:
Device: Flow Diverter (Tonbridge) — The device is a self-expanding vascular stent system, which consists of a stent and a delivery system. The stent is made of platinum core nickel-titanium alloy material. The delivery system is composed of a delivery guide wire and an introducer sheath. The stent and the delivery guide wire are pre-installed in the introducer sheath.

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of the Flow Diverter (Tonbridge) by collecting data from subjects who receive endovascular treatment of intracranial aneurysms.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm clinical trial carried out in 7 research centers over China. In this study, enrolled patients are treated with the Flow Diverter (Tonbridge) for intracranial aneurysms. The objective of this study is to evaluate the effectiveness and safety of the Flow Diverter (Tonbridge) for treatment of intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years, any gender;
* A single unruptured intracranial aneurysm locates in the intracranial segment of internal carotid artery (ICA) or vertebral artery (VA), which diagnosed by DSA;
* The maximal diameter of the target aneurysm < 10 mm diagnosed by DSA;
* The target aneurysm with a neck ≥ 4 mm or a dome to neck ratio < 2 diagnosed by DSA;
* The target aneurysm with a parent vessel diameter of 2.0-6.5 mm;
* Subject or guardian is able to understand the purpose of study, shows sufficient compliance with the study protocol and provides a signed informed consent form.

Exclusion Criteria:

* Diagnosed as with cerebrovascular malformations;
* Intracranial hemorrhage within 30 days pre-procedure;
* Modified Rankin Scale (mRS) score ≥ 3 in pre-procedure;
* Platelet (PLT) < 60×10^9/L or known platelet dysfunction or International Normalized Ratio (INR) > 1.5;
* Heart, lung, liver and renal failure or other severe diseases (such as intracranial tumor, systemic infection, disseminated intravascular coagulation, myocardial infarction within 12 months before enrollment, history of severe psychosis, severe stenosis or occlusion of cerebral feeding artery);
* Subject who is not appropriate for flow diverter delivery and deployment judged by investigators (severe stenosis of parent artery, severe tortuosity of parent artery, stent failing to reach the lesion, stent in the target lesion of parent artery, etc.);
* Major surgery within 30 days before enrollment, or intending to receive surgery within 180 days after enrollment;
* Allergic history of anesthetics and contrast agents, or contraindication for dual antiplatelet or/and anticoagulant therapy;
* Allergic history of metals such as nickel-titanium alloy;
* Life expectancy < 12 months;
* Pregnant or breastfeeding women;
* Subject has participated in other drug or medical device clinical trials within 1 month before signing informed consent;
* Other conditions judged by the investigators as unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Complete occlusion rate of aneurysms at 12 months | 360±30 days post-procedure
  Complete occlusion is defined as no contrast agent in the aneurysm (Raymond-Roy class I) which is diagnosed by cerebrovascular DSA at 12 months post-procedure.

SECONDARY OUTCOMES:
Immediate procedural success rate | intra-procedure
  Intraoperative cerebrovascular DSA is performed to determine whether the investigational device positions exactly and covers the aneurysm neck effectively.
Complete occlusion rate of aneurysms at 6 months | 180±30 days post-procedure
  Complete occlusion is defined as no contrast agent in the aneurysm (Raymond-Roy class I) which is diagnosed by MRA/CTA at 6 months post-procedure.
Successful occlusion rate of aneurysms at 12 months | 360±30 days post-procedure
  Successful occlusion is defined as Raymond-Roy class I or II, which is diagnosed by DSA at 12 months post-procedure.
Incidence of new-onset stroke in the territory supplied by the treated artery or neurologic death at 12 months | 360±30 days post-procedure
  New-onset stroke is defined as the occurrence of new stroke with an increase of ≥ 4 points in the subjects' NIHSS score from preoperative baseline. Neurologic death is defined as death due to neurologic reasons directly.
Incidence of technical complications | intra-procedure
  Technical complications include but not limited to: stent incomplete opening, stent migration, stent herniation into the aneurysm sac, in-stent thrombosis, operation injury, etc.
Incidence of any stroke | 30±7 days, 360±30 days post-procedure
  Stroke includes hemorrhagic stroke and symptomatic ischemic stroke.
Incidence of parent artery stenosis ( > 50%）in target area at 12 months | 360±30 days post-procedure
  Parent artery stenosis in target area is defined as stenosis degree > 50%. Using postoperative cerebrovascular DSA at 12 months is performed to determine.
Incidence of parent artery occlusion in target area at 12 months | 360±30 days post-procedure
  Postoperative cerebrovascular DSA at 12 months is performed to determine whether parent artery in target area is occluded.
Incidence of adverse events | pre-procedure, intra-procedure, within 24 hours, 30±7 days, 90±14 days, 180±30 days, 360±30 days post-procedure
  "Incidence of adverse events" is the proportion of subjects with adverse events using the investigational device.
Incidence of serious adverse events | pre-procedure, intra-procedure, within 24 hours, 30±7 days, 90±14 days, 180±30 days, 360±30 days post-procedure
  "Incidence of serious adverse events" is the proportion of subjects with serious adverse events using the investigational device.
Mortality rate | 30±7 days, 360±30 days post-procedure
  Deaths due to any cause are calculated.
Operation satisfaction rate | intra-procedure
  The 5-point Likert scale is used to evaluate the operation satisfaction from three aspects: push performance, retracting performance and release performance. "Operation satisfaction rate" is defined as the proportion of investigational devices with Likert score ≥ 12 points.
Incidence of device deficiency | intra-procedure, 360±30 days post-procedure
  Device deficiency is the unreasonable risk that may endanger human health and life safety in the normal use of medical devices during clinical trials, such as labeling errors, quality problems, malfunctions, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital
Locations (7):
- China (7):
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Xinqiao Hospital, Army Medical University, Chongqing
  - Changhai Hospital of Shanghai, Shanghai
  - Huashan Hospital Fudan University, Shanghai